CLINICAL TRIAL: NCT02837497
Title: Improving Outcomes After Pediatric Cardiac Arrest
Brief Title: The ICU-Resuscitation Project (ICU-RESUS)
Acronym: ICU-RESUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Utah (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 15-012576; R01HL131544 (NIH); UG1HD063108 (NIH)
Record Dates: First submitted 2016-07-14; First posted 2016-07-19 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Cardiac Arrest
Keywords: pediatric; heart arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard ICU resuscitation practices
- ICU-RESUS CPR Improvement Bundle (Experimental): ICU-RESUS bundle implementation: 1) point-of-care bedside CPR training; and 2) post-cardiac arrest debriefings.
  Interventions: Other: ICU-RESUS CPR Improvement Bundle

INTERVENTIONS:
Other: ICU-RESUS CPR Improvement Bundle — 1. Point-of-care CPR training
  2. Post-cardiac arrest educational debriefings
  Other Names: ICU-RESUS
  Arms: ICU-RESUS CPR Improvement Bundle

SUMMARY:
Pediatric cardiac arrest affects thousands of hospitalized children each year. High quality cardiopulmonary resuscitation (CPR) saves lives, but is difficult to achieve. The objective of this study is to determine if a novel patient-centric resuscitation care improvement bundle consisting of bedside CPR training and multidisciplinary reviews of each cardiac arrest improves CPR quality and survival outcomes in a multi-center trial.

DETAILED DESCRIPTION:
Pediatric cardiac arrest affects thousands of hospitalized children each year. Progressive heart and lung failure is a predisposing cause in the majority of these events. While cardiac arrest survival outcomes have improved over the last decade, more than half of these children will not live to hospital discharge. As brain injury complicates care in those who do survive, the burden to these children and the public's health is substantial.

Cardiopulmonary resuscitation (CPR) - the medical procedure of providing chest compressions and ventilations during cardiac arrest - is life saving, and higher quality CPR is more effective at doing so. However, providing high quality care during the resuscitation of a child is difficult. Attempts to improve care through conventional training methods have not been successful; therefore, interventions to improve the quality of pediatric CPR and outcomes are needed.

The objective of this study is to determine if a novel resuscitation care improvement bundle that improved outcomes in a single center intensive care unit (ICU) efficacy study is generalizable to other pediatric institutions in a multi-center effectiveness trial. The ICU-Resuscitation (ICU-RESUS) bundle includes: 1) CPR training at the point-of-care (in the ICU rather than a classroom away from patients); and 2) interdisciplinary structured reviews of each cardiac arrest that emphasize patient-centric physiology intended to optimize intra-arrest and post-arrest care. The ICU-RESUS bundle substantially improved CPR quality and nearly doubled the number of children surviving their event during the single center efficacy trial. In this study, a multi-institutional parallel stepped-wedge hybrid cluster-randomized trial, which leverages the existing infrastructure of the National Institute of Child Health and Human Development (NICHD)-funded Collaborative Pediatric Critical Care Research Network (CPCCRN), is proposed with the following aims: 1) Evaluate the effectiveness of the ICU-RESUS interventional bundle to improve outcomes of children treated for an ICU cardiac arrest; and 2) Evaluate the effectiveness of the ICU-RESUS interventional bundle to improve the quality of CPR provided by ICU healthcare providers in the population of children treated for an ICU cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 37 weeks and less than or equal to18 years of age;
* AND Received CPR in the ICU setting

Exclusion Criteria:

* Pre-existing terminal illness and patient not expected to survive to hospital discharge.
* Lack of commitment to aggressive ICU therapies.
* Brain death determination prior to CPR event.
* First CPR event associated with this hospital admission was an out-of-hospital CPR event.

Ages: 37 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1127 (Actual)
Dates: Start 2016-10; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Good neurological survival | Baseline and hospital discharge
  Pediatric cerebral performance category of less than or equal to 3 or no change from baseline.

SECONDARY OUTCOMES:
Excellent CPR | During cardiopulmonary resuscitation
  A composite variable of systolic blood pressure >60 mmHg for neonates, >80 mmHg for infants, or >100 mmHg for older patients AND compression rate between 100-120 / minute, AND a chest compression fraction greater than or equal to 80%.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sutton, MD MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Berg RA, Nadkarni VM, Clark AE, Moler F, Meert K, Harrison RE, Newth CJ, Sutton RM, Wessel DL, Berger JT, Carcillo J, Dalton H, Heidemann S, Shanley TP, Zuppa AF, Doctor A, Tamburro RF, Jenkins TL, Dean JM, Holubkov R, Pollack MM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network. Incidence and Outcomes of Cardiopulmonary Resuscitation in PICUs. Crit Care Med. 2016 Apr;44(4):798-808. doi: 10.1097/CCM.0000000000001484. PMID 26646466
- [Background] Wolfe H, Maltese MR, Niles DE, Fischman E, Legkobitova V, Leffelman J, Berg RA, Nadkarni VM, Sutton RM. Blood Pressure Directed Booster Trainings Improve Intensive Care Unit Provider Retention of Excellent Cardiopulmonary Resuscitation Skills. Pediatr Emerg Care. 2015 Nov;31(11):743-7. doi: 10.1097/PEC.0000000000000394. PMID 25822236
- [Background] Sutton RM, Friess SH, Naim MY, Lampe JW, Bratinov G, Weiland TR 3rd, Garuccio M, Nadkarni VM, Becker LB, Berg RA. Patient-centric blood pressure-targeted cardiopulmonary resuscitation improves survival from cardiac arrest. Am J Respir Crit Care Med. 2014 Dec 1;190(11):1255-62. doi: 10.1164/rccm.201407-1343OC. PMID 25321490
- [Background] Sutton RM, French B, Niles DE, Donoghue A, Topjian AA, Nishisaki A, Leffelman J, Wolfe H, Berg RA, Nadkarni VM, Meaney PA. 2010 American Heart Association recommended compression depths during pediatric in-hospital resuscitations are associated with survival. Resuscitation. 2014 Sep;85(9):1179-84. doi: 10.1016/j.resuscitation.2014.05.007. Epub 2014 May 16. PMID 24842846
- [Background] Wolfe H, Zebuhr C, Topjian AA, Nishisaki A, Niles DE, Meaney PA, Boyle L, Giordano RT, Davis D, Priestley M, Apkon M, Berg RA, Nadkarni VM, Sutton RM. Interdisciplinary ICU cardiac arrest debriefing improves survival outcomes*. Crit Care Med. 2014 Jul;42(7):1688-95. doi: 10.1097/CCM.0000000000000327. PMID 24717462
- [Background] Topjian AA, French B, Sutton RM, Conlon T, Nadkarni VM, Moler FW, Dean JM, Berg RA. Early postresuscitation hypotension is associated with increased mortality following pediatric cardiac arrest. Crit Care Med. 2014 Jun;42(6):1518-23. doi: 10.1097/CCM.0000000000000216. PMID 24561563
- [Derived] Ullman NL, Reeder RW, Topjian A, Morgan RW, Berg RA, Nadkarni VM, Palmer CA, Sutton RM, Press CA, Kirschen MP; ICU-RESUS, CPCCRN Investigators. Severe intracranial hemorrhage or ischemia associated with unfavorable outcomes after pediatric in-hospital cardiac arrest. Resuscitation. 2026 Jan;218:110886. doi: 10.1016/j.resuscitation.2025.110886. Epub 2025 Nov 7. PMID 41207462
- [Derived] Morgan RW, Reeder RW, Carcillo JA, Carpenter TC, Fitzgerald JC, Graham K, Kilbaugh TJ, Meert KL, Nadkarni VM, Palmer CA, Sharron MP, Weiss SL, Wolfe HA, Ahmed T, Bell MJ, Bishop R, Burns C, Diddle JW, Fink EL, Franzon D, Frazier AH, Friess SH, Hehir DA, Horvat CM, Huard LL, Maa T, McQuillen PS, Mourani PM, Naim MY, Pollack MM, Sapru A, Srivastava N, Yates AR, Berg RA, Sutton RM; for the ICU-Resuscitation Project (ICU-RESUS) Investigators and the Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network Investigators. Outcomes, Characteristics, and Physiology of In-Hospital Cardiac Arrest in Children With Sepsis. Crit Care Med. 2025 Aug 1;53(8):e1529-e1541. doi: 10.1097/CCM.0000000000006739. Epub 2025 Jun 25. PMID 40558671
- [Derived] Siems A, Naim MY, Berg RA, Reeder RW, Ahmed T, Bell MJ, Bishop R, Bochkoris M, Burns C, Carcillo JA, Carpenter TC, Diddle JW, Federman M, Fernandez R, Fink EL, Franzon D, Frazier AH, Friess SH, Graham K, Hall M, Harding ML, Hehir DA, Horvat CM, Huard LL, Kilbaugh TJ, Maa T, Manga A, McQuillen PS, Meert KL, Mourani PM, Nadkarni VM, Notterman D, Pollack MM, Qunibi DW, Sapru A, Schneiter C, Sharron MP, Srivastava N, Tabbutt S, Tilford B, Viteri S, Wessel D, Wolfe HA, Yates AR, Zuppa AF, Morgan RW, Sutton RM. Association of Early Epinephrine with Hemodynamics and Outcome in Pediatric In-Hospital Cardiac Arrest: A Secondary Analysis of a Multicenter, Cluster-randomized Clinical Trial Intensive Care Unit Resuscitation (ICU-RESUS). Ann Am Thorac Soc. 2025 Sep;22(9):1361-1371. doi: 10.1513/AnnalsATS.202408-825OC. PMID 40466056
- [Derived] Kirschen MP, Ullman NL, Reeder RW, Ahmed T, Bell MJ, Berg RA, Burns C, Carcillo JA, Carpenter TC, Wesley Diddle J, Federman M, Fink EL, Frazier AH, Friess SH, Graham K, Horvat CM, Huard LL, Kilbaugh TJ, Maa T, Manga A, McQuillen PS, Meert KL, Morgan RW, Mourani PM, Nadkarni VM, Naim MY, Notterman D, Palmer CA, Pollack MM, Sapru A, Sharron MP, Srivastava N, Tilford B, Viteri S, Wolfe HA, Yates AR, Topjian A, Sutton RM, Press CA. Practice patterns for acquiring neuroimaging after pediatric in-hospital cardiac arrest. Resuscitation. 2025 Feb;207:110506. doi: 10.1016/j.resuscitation.2025.110506. Epub 2025 Jan 21. PMID 39848427
- [Derived] Nishisaki A, Reeder RW, McGovern EL, Ahmed T, Bell MJ, Bishop R, Bochkoris M, Burns C, Carcillo JA, Carpenter TC, Diddle W, Federman M, Fink EL, Franzon D, Frazier AH, Friess SH, Graham K, Hall M, Hehir DA, Horvat CM, Huard LL, Maa T, Manga A, McQuillen P, Meert KL, Morgan RW, Mourani PM, Nadkarni VM, Naim MY, Notterman D, Palmer CA, Sapru A, Schneiter C, Sharron MP, Srivastava N, Viteri S, Wessel D, Wolfe HA, Yates AR, Zuppa AF, Sutton RM, Berg RA. Brief report: incidence and outcomes of pediatric tracheal intubation-associated cardiac arrests in the ICU-RESUS clinical trial. Crit Care. 2024 Aug 30;28(1):286. doi: 10.1186/s13054-024-05065-0. PMID 39215367
- [Derived] Yates AR, Naim MY, Reeder RW, Ahmed T, Banks RK, Bell MJ, Berg RA, Bishop R, Bochkoris M, Burns C, Carcillo JA, Carpenter TC, Dean JM, Diddle JW, Federman M, Fernandez R, Fink EL, Franzon D, Frazier AH, Friess SH, Graham K, Hall M, Hehir DA, Horvat CM, Huard LL, Maa T, Manga A, McQuillen PS, Morgan RW, Mourani PM, Nadkarni VM, Notterman D, Pollack MM, Sapru A, Schneiter C, Sharron MP, Srivastava N, Tilford B, Viteri S, Wessel D, Wolfe HA, Yeh J, Zuppa AF, Sutton RM, Meert KL. Early Cardiac Arrest Hemodynamics, End-Tidal C o2 , and Outcome in Pediatric Extracorporeal Cardiopulmonary Resuscitation: Secondary Analysis of the ICU-RESUScitation Project Dataset (2016-2021). Pediatr Crit Care Med. 2024 Apr 1;25(4):312-322. doi: 10.1097/PCC.0000000000003423. Epub 2023 Dec 13. PMID 38088765
- [Derived] Morgan RW, Reeder RW, Bender D, Cooper KK, Friess SH, Graham K, Meert KL, Mourani PM, Murray R, Nadkarni VM, Nataraj C, Palmer CA, Srivastava N, Tilford B, Wolfe HA, Yates AR, Berg RA, Sutton RM; ICU-RESUS and Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network (CPCCRN) Investigator Groups. Associations Between End-Tidal Carbon Dioxide During Pediatric Cardiopulmonary Resuscitation, Cardiopulmonary Resuscitation Quality, and Survival. Circulation. 2024 Jan 30;149(5):367-378. doi: 10.1161/CIRCULATIONAHA.123.066659. Epub 2023 Nov 6. PMID 37929615
- [Derived] Gardner MM, Hehir DA, Reeder RW, Ahmed T, Bell MJ, Berg RA, Bishop R, Bochkoris M, Burns C, Carcillo JA, Carpenter TC, Dean JM, Diddle JW, Federman M, Fernandez R, Fink EL, Franzon D, Frazier AH, Friess SH, Graham K, Hall M, Harding ML, Horvat CM, Huard LL, Maa T, Manga A, McQuillen PS, Meert KL, Morgan RW, Mourani PM, Nadkarni VM, Naim MY, Notterman D, Pollack MM, Sapru A, Schneiter C, Sharron MP, Srivastava N, Tilford B, Viteri S, Wessel D, Wolfe HA, Yates AR, Zuppa AF, Sutton RM, Topjian AA. Identification of post-cardiac arrest blood pressure thresholds associated with outcomes in children: an ICU-Resuscitation study. Crit Care. 2023 Oct 7;27(1):388. doi: 10.1186/s13054-023-04662-9. PMID 37805481
- [Derived] Federman M, Sutton RM, Reeder RW, Ahmed T, Bell MJ, Berg RA, Bishop R, Bochkoris M, Burns C, Carcillo JA, Carpenter TC, Dean JM, Diddle JW, Fernandez R, Fink EL, Franzon D, Frazier AH, Friess SH, Graham K, Hall M, Hehir DA, Horvat CM, Huard LL, Kirkpatrick T, Maa T, Maitoza LA, Manga A, McQuillen PS, Meert KL, Morgan RW, Mourani PM, Nadkarni VM, Notterman D, Palmer CA, Pollack MM, Sapru A, Schneiter C, Sharron MP, Srivastava N, Tilford B, Viteri S, Wessel D, Wolfe HA, Yates AR, Zuppa AF, Naim MY. Survival With Favorable Neurologic Outcome and Quality of Cardiopulmonary Resuscitation Following In-Hospital Cardiac Arrest in Children With Cardiac Disease Compared With Noncardiac Disease. Pediatr Crit Care Med. 2024 Jan 1;25(1):4-14. doi: 10.1097/PCC.0000000000003368. Epub 2023 Sep 7. PMID 37678381
- [Derived] Morgan RW, Reeder RW, Ahmed T, Bell MJ, Berger JT, Bishop R, Bochkoris M, Burns C, Carcillo JA, Carpenter TC, Dean JM, Diddle JW, Federman M, Fernandez R, Fink EL, Franzon D, Frazier AH, Friess SH, Graham K, Hall M, Hehir DA, Himebauch AS, Horvat CM, Huard LL, Maa T, Manga A, McQuillen PS, Meert KL, Mourani PM, Nadkarni VM, Naim MY, Notterman D, Page K, Pollack MM, Sapru A, Schneiter C, Sharron MP, Srivastava N, Tabbutt S, Tilford B, Viteri S, Wessel D, Wolfe HA, Yates AR, Zuppa AF, Berg RA, Sutton RM. Outcomes and characteristics of cardiac arrest in children with pulmonary hypertension: A secondary analysis of the ICU-RESUS clinical trial. Resuscitation. 2023 Sep;190:109897. doi: 10.1016/j.resuscitation.2023.109897. Epub 2023 Jul 3. PMID 37406760
- [Derived] Cashen K, Reeder RW, Ahmed T, Bell MJ, Berg RA, Burns C, Carcillo JA, Carpenter TC, Dean JM, Diddle JW, Federman M, Fink EL, Frazier AH, Friess SH, Graham K, Hall M, Hehir DA, Horvat CM, Huard LL, Maa T, Manga A, McQuillen PS, Morgan RW, Mourani PM, Nadkarni VM, Naim MY, Notterman D, Palmer CA, Pollack MM, Schneiter C, Sharron MP, Srivastava N, Wessel D, Wolfe HA, Yates AR, Zuppa AF, Sutton RM, Meert KL; for the Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network (CPCCRN) and National Heart Lung and Blood Institute ICU-RESUScitation Project Investigators. Sodium Bicarbonate Use During Pediatric Cardiopulmonary Resuscitation: A Secondary Analysis of the ICU-RESUScitation Project Trial. Pediatr Crit Care Med. 2022 Oct 1;23(10):784-792. doi: 10.1097/PCC.0000000000003045. Epub 2022 Jul 26. PMID 35880872
- [Derived] ICU-RESUS and Eunice Kennedy Shriver National Institute of Child Health; Human Development Collaborative Pediatric Critical Care Research Network Investigator Groups; Sutton RM, Wolfe HA, Reeder RW, Ahmed T, Bishop R, Bochkoris M, Burns C, Diddle JW, Federman M, Fernandez R, Franzon D, Frazier AH, Friess SH, Graham K, Hehir D, Horvat CM, Huard LL, Landis WP, Maa T, Manga A, Morgan RW, Nadkarni VM, Naim MY, Palmer CA, Schneiter C, Sharron MP, Siems A, Srivastava N, Tabbutt S, Tilford B, Viteri S, Berg RA, Bell MJ, Carcillo JA, Carpenter TC, Dean JM, Fink EL, Hall M, McQuillen PS, Meert KL, Mourani PM, Notterman D, Pollack MM, Sapru A, Wessel D, Yates AR, Zuppa AF. Effect of Physiologic Point-of-Care Cardiopulmonary Resuscitation Training on Survival With Favorable Neurologic Outcome in Cardiac Arrest in Pediatric ICUs: A Randomized Clinical Trial. JAMA. 2022 Mar 8;327(10):934-945. doi: 10.1001/jama.2022.1738. PMID 35258533
- [Derived] Reeder RW, Girling A, Wolfe H, Holubkov R, Berg RA, Naim MY, Meert KL, Tilford B, Carcillo JA, Hamilton M, Bochkoris M, Hall M, Maa T, Yates AR, Sapru A, Kelly R, Federman M, Michael Dean J, McQuillen PS, Franzon D, Pollack MM, Siems A, Diddle J, Wessel DL, Mourani PM, Zebuhr C, Bishop R, Friess S, Burns C, Viteri S, Hehir DA, Whitney Coleman R, Jenkins TL, Notterman DA, Tamburro RF, Sutton RM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network (CPCCRN). Improving outcomes after pediatric cardiac arrest - the ICU-Resuscitation Project: study protocol for a randomized controlled trial. Trials. 2018 Apr 3;19(1):213. doi: 10.1186/s13063-018-2590-y. PMID 29615134